CLINICAL TRIAL: NCT03726333
Title: A PHASE 1 STUDY TO EVALUATE THE EFFECT OF HEPATIC IMPAIRMENT ON THE PHARMACOKINETICS AND SAFETY OF LORLATINIB IN ADVANCED CANCER PATIENTS
Brief Title: Hepatic Impairment Study for Lorlatinib in Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study stopped due to lack of enrollment
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B7461009; lorlatinib HEPATIC IMPAIRMENT (Other: Alias Study Number); HEPATIC IMPAIRMENT (Other: Alias Study Number)
Record Dates: First submitted 2018-09-24; First posted 2018-10-31 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-01

CONDITIONS: Advanced Cancers
Keywords: hepatic impairment; lorlatinib; cancer; pharmacokinetic; Lung cancer
MeSH Terms: conditions — Neoplasms; Lung Neoplasms | interventions — lorlatinib

STUDY DESIGN:
Intervention Model Description: Patients in the study will be assigned to different groups according to their liver function. Patients in each group will receive specific lorlatinib dose. Plasma samples for pharmacokinetic analysis will be collected in all patients. Safety and efficacy will also be followed in all patients until at least 28 days after the last study treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group A1 Normal hepatic function (Active Comparator): continued daily administration of lorlatinib in patients with normal hepatic function
  Interventions: Drug: lorlatinib
- Group A2 Normal hepatic function (Active Comparator): continued daily administration of lorlatinib in patients with normal hepatic function
  Interventions: Drug: lorlatinib
- Group B mild hepatic impairment (Experimental): continued daily administration of lorlatinib in patients with mild hepatic impairment
  Interventions: Drug: lorlatinib
- Group C moderate hepatic impairment (Experimental): continued daily administration of lorlatinib in patients with moderate hepatic impairment
  Interventions: Drug: lorlatinib
- Group D severe hepatic impairment (Experimental): continued daily administration of lorlatinib in patients with severe hepatic impairment
  Interventions: Drug: lorlatinib

INTERVENTIONS:
Drug: lorlatinib — continued daily administration of 100 mg lorlatinib
  Arms: Group A1 Normal hepatic function
Drug: lorlatinib — continued daily administration of lorlatinib at the dose level same as Group C for the first 22 days and 100 mg QD afterwards
  Arms: Group A2 Normal hepatic function
Drug: lorlatinib — continued daily administration of 100 mg QD lorlatinib
  Arms: Group B mild hepatic impairment
Drug: lorlatinib — continued daily administration of lorlatinib at 50 mg QD initially and may be adjusted based on PK and safety results from the initial several patients
  Arms: Group C moderate hepatic impairment
Drug: lorlatinib — continued daily administration of lorlatinib at the dose level determined based on preliminary PK and safety results from first several patients in Group C
  Arms: Group D severe hepatic impairment

SUMMARY:
This is a phase 1 study in advanced cancer patients with varied hepatic functions to evaluate the potential effect of hepatic impairment on pharmacokinetics and safety of lorlatinib and provide dose recommendation for patients with hepatic impairment if possible.

DETAILED DESCRIPTION:
This will be a Phase 1, open label, multi center, multiple dose, non randomized, Phase 1 clinical trial of lorlatinib in advanced cancer patients with varying degrees of hepatic impairment and necessary age , weight , and gender matched prospect normal hepatic function patients. This study is intended to evaluate the potential effect of hepatic impairments on the PK and safety of lorlatinib after daily administration of lorlatinib and to provide dosing recommendation for patients with varied degree of hepatic impairment if possible.

Patients in the study will be assigned to different groups (A1, normal liver function, control for group B; A2, normal liver function, control for group C; B, mild hepatic impairment; C, moderate hepatic impairment; D, severe hepatic impairment) according to their liver function. The enrollment of approximately 76 advanced cancer patients is anticipated in this study in order to have 8 PK-evaluable patients in each of Groups A1, A2, B and C, and 6 PK-evaluable patients in Group D for final statistical analysis. Evaluable patients are those who complete the planned PK sample collection on Cycle 2 Day 1 and have no lorlatinib dose modification until completion of Cycle 2 Day 1 PK evaluation. Patients who are not evaluable for PK will be replaced. Each patient will be treated with repeated oral once daily doses of lorlatinib in 21-day cycles until disease progression, patient refusal, or unacceptable toxicity occurs. The dose schedule may be modified as necessary for individual patients according to tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid malignancy or lymphoma that is metastatic or unresectable, and for which standard curative or palliative measures do not exist, or are no longer effective;
* Biliary obstruction with a biliary drain or stent;
* Neurologically stable gliomas and brain metastases;
* ECOG performance status of 0, 1, or 2;
* adequate bone marrow function;
* adequate pancreatic function;
* adequate renal function;
* female patients with negative pregnancy test

Exclusion Criteria:

* untreated esophageal varices; uncontrolled ascites;
* episodes of hepatic encephalopathy within the last 4 weeks;
* spinal cord compression; major surgery within 4 weeks prior to enrollment;
* radiation therapy within 2 weeks prior to enrollment;
* last anti-cancer treatment within 2 weeks prior to screening;
* previous high-dose chemotherapy requiring stem cell rescue;
* prior to irradiation to >25% of the bone marrow;
* gastrointestinal abnormalities;
* known prior or suspected hypersensitivity to lorlatinib or lorlatinib tablet;
* clinically significant bacterial, fungal or viral infections for non-liver cancer patients;
* clinically significant cardiovascular disease;
* uncontrolled hypertension; acute pancreatitis with predisposing characteristics;
* history of grade 3 or 4 interstitial fibrosis or interstitial lung disease;
* active hemoelysis or evidence of biliary sepsis;
* prior major gastrointestinal surgery;
* concurrent use of known strong CYP3A inhibitors, inducers and P-gp substrates with a narrow therapeutic index;
* concurrent use of CYP3A substrates with narrow therapeutic indices;
* prior treatment with lorlatinib; active bleeding disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (10):
  - University of Colorado Denver CTO (CTRC), Aurora, Colorado
  - University of Colorado Hospital, Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - University of Colorado Hospital, Anschutz Inpatient Pavilion (AIP), Aurora, Colorado
  - University of Colorado Hospital, Anschutz Outpatient Pavilion (AOP), Aurora, Colorado
  - Emory University Hospital, Atlanta, Georgia
  - Investigational Drug Service, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Mays Cancer Center, San Antonio, Texas
  - University Health System, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461009

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 4 participants were screened. Among them, 1 participant was enrolled and treated in Group B (mild impairment), 1 participant was eligible for Group A (normal) but not enrolled as Group A was not open for enrolment at that time, and 2 participants were screen failed.
Groups:
- Group A1 Normal Hepatic Function: Continued daily administration of lorlatinib 100 mg in patients with normal hepatic function until disease progression, patient refusal, or unacceptable toxicity occurrence
- Group A2 Normal Hepatic Function: Continued daily administration of lorlatinib in patients with normal hepatic function at the dose level same as Group C for the first 22 days and 100 mg once a day (QD) afterwards.
- Group B Mild Hepatic Impairment: Continued daily administration of lorlatinib in patients with mild hepatic impairment. The participant received lorlatinib 100 mg QD in Cycle 1 and lorlatinib 75 mg QD in Cycle 2.
- Group C Moderate Hepatic Impairment: Continued daily administration of lorlatinib in patients with moderate hepatic impairment at 50 mg QD initially and may be adjusted based on PK and safety results from the initial several patients.
- Group D Severe Hepatic Impairment: Continued daily administration of lorlatinib in patients with severe hepatic impairment at the dose level determined based on preliminary PK and safety results from first several patients in Group C.
Period: Overall Study
Arm/Group | Group A1 Normal Hepatic Function | Group A2 Normal Hepatic Function | Group B Mild Hepatic Impairment | Group C Moderate Hepatic Impairment | Group D Severe Hepatic Impairment
Started | 0 | 0 | 1 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — Data cannot be reported because doing so would risk re-identification of participants.
  Between 18 and 65 years | NA — Data cannot be reported because doing so would risk re-identification of participants.
  >=65 years | NA — Data cannot be reported because doing so would risk re-identification of participants.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Data cannot be reported because doing so would risk re-identification of the participant.
  Male | NA — Data cannot be reported because doing so would risk re-identification of the participant..
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | NA — Data cannot be reported because doing so would risk re-identification of participants.
  Not Hispanic or Latino | NA — Data cannot be reported because doing so would risk re-identification of participants.
  Unknown or Not Reported | NA — Data cannot be reported because doing so would risk re-identification of participants.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Data cannot be reported because doing so would risk re-identification of participants.
  Asian | NA — Data cannot be reported because doing so would risk re-identification of participants.
  Native Hawaiian or Other Pacific Islander | NA — Data cannot be reported because doing so would risk re-identification of participants.
  Black or African American | NA — Data cannot be reported because doing so would risk re-identification of participants.
  White | NA — Data cannot be reported because doing so would risk re-identification of participants.
  More than one race | NA — Data cannot be reported because doing so would risk re-identification of participants.
  Unknown or Not Reported | NA — Data cannot be reported because doing so would risk re-identification of participants.

OUTCOME MEASURES:

1. Primary Outcome: Area Under Plasma Lorlatinib Concentration-Time Curve From Time 0 to Dosing Interval of 24 Hours (AUC24) at Steady State On Cycle 2 Day 1
Description: AUC24 was defined as area under the plasma concentration time profile during 1 dosing interval (24 hours).
Time Frame: Cycle 2 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: The analysis population included all enrolled participants who received at least 1 dose of lorlatinib and had sufficient information to estimate at least 1 of the pharmacokinetic parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
nanogram*hour per milliliter (ng*hr/mL) | NA (NA) — No PK parameter estimation was performed for the 1 treated participant

2. Primary Outcome: Observed Maximal Plasma Concentration (Cmax) at Steady State on Cycle 2 Day 1
Description: Cmax was defined as maximum plasma concentration and was observed directly from data.
Time Frame: Cycle 2 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
nanogram per milliliter (ng/mL) | NA (NA) — No PK parameter estimation was performed for the 1 treated participant.

3. Secondary Outcome: Number Of Patients Experienced Treatment Emergent Adverse Event Assessed by Investigator
Description: An Adverse event (AE) was any untoward medical occurrence in a participant. A serious AE was any untoward medical occurrence at any dose that resulted in death; was life-threatening; required hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect or that was considered to be an important medical event. AEs were graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. The grades were defined as follows: Grade 0: no change from normal or reference range; Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death related to AE. The focus of AE summaries was on treatment-emergent AE (TEAE). An AE was considered TEAE if the event occurred during the on-treatment period.
Time Frame: From Screening (within 28 days prior to Cycle 1 Day 1) through and including at least 28 days after after the last lorlatinib dose. The duration is approximately 42 days.
Population: The analysis population included all enrolled participants who received at least 1 dose of lorlatinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
Participants
  All-causality TEAEs | NA — Data cannot be reported because doing so would risk re-identification of the participant.
  Treatment-related TEAEs | NA — Data cannot be reported because doing so would risk re-identification of the participant.
  All-causality serious AEs | NA — Data cannot be reported because doing so would risk re-identification of the participant.
  Treatment-related serious AEs | NA — Data cannot be reported because doing so would risk re-identification of the participant.
  All-causalities AEs ≥Grade 3 | NA — Data cannot be reported because doing so would risk re-identification of the participant.
  Treatment-related AEs ≥Grade 3 | NA — Data cannot be reported because doing so would risk re-identification of the participant.
  All-causalities Grade 1 AEs | NA — Data cannot be reported because doing so would risk re-identification of the participant.
  Treatment-related Grade 1 AEs | NA — Data cannot be reported because doing so would risk re-identification of the participant.
  All-causalities Grade 2 AEs | NA — Data cannot be reported because doing so would risk re-identification of the participant.
  Treatment-related Grade 2 AEs | NA — Data cannot be reported because doing so would risk re-identification of the participant.

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a best overall confirmed response of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1 relative to the response-evaluable population.
Time Frame: Baseline up to approximately 1 year
Population: The analysis population included all enrolled participants who received at least 1 dose of lorlatinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
Percentage of participants | 0 [0 to 97.5]

5. Secondary Outcome: Duration of Response (DR)
Description: DR was measured from the date that an objective tumor response (CR or PR) was first documented (whichever occurred first) to date of objective tumor progression or death due to any cause, whichever occurred first.
Time Frame: Baseline up to approximately 1 year
Population: The analysis population included all enrolled participants who received at least 1 dose of lorlatinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
Months | NA [NA to NA] — The participant had an overall objective tumor assessment of progressive disease. As no patient responded DR is Not Applicable.

6. Secondary Outcome: Lorlatinib Area Under Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) After Single Dose on Cycle 1 Day 1
Description: AUClast was defined as area under the plasma concentration time profile from time 0 to the time of the last quantifiable concentration (Clast)
Time Frame: Cycle 1 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
ng*hr/mL | NA (NA) — No PK parameter estimation was performed for the 1 treated participant

7. Secondary Outcome: The Time of The Last Quantifiable Concentration (Tlast) of Lorlatinib After Single Dose on Cycle 1 Day 1
Description: Tlast was defined as the time of the last quantifiable concentration.
Time Frame: Cycle 1 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
hour | NA [NA to NA] — No PK parameter estimation was performed for the 1 treated participant

8. Secondary Outcome: The Time to Cmax (Tmax) of Lorlatinib After Single Dose on Cycle 1 Day 1
Description: Tmax was defined as time for Cmax.
Time Frame: Cycle 1 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
hour | NA [NA to NA] — No PK parameter estimation was performed for the 1 treated participant

9. Secondary Outcome: Observed Minimal Plasma Concentration (Cmin) at Steady State On Cycle 2 Day 1
Description: Cmin was defined as minimum plasma concentration and was observed directly from data.
Time Frame: Cycle 2 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
ng/mL | NA (NA) — No PK parameter estimation was performed for the 1 treated participant.

10. Secondary Outcome: Plasma Lorlatinib AUClast at Steady State On Cycle 2 Day 1
Description: AUClast was defined as area under the plasma concentration time profile from time 0 to the time of Clast.
Time Frame: Cycle 2 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
ng*hr/mL | NA (NA) — No PK parameter estimation was performed for the 1 treated participant.

11. Secondary Outcome: Plasma Lorlatinib Tlast at Steady State On Cycle 2 Day 1
Description: Tlast was defined as the time of the last quantifiable concentration.
Time Frame: Cycle 2 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
hour | NA [NA to NA] — No PK parameter estimation was performed for the 1 treated participant

12. Secondary Outcome: Apparent Clearance (CL/F) at Steady State On Cycle 2 Day 1
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CL/F was calculated as Dose/AUC24 at steady-state.
Time Frame: Cycle 2 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
Liter per hour (L/hr) | NA (NA) — No PK parameter estimation was performed for the 1 treated participant.

13. Secondary Outcome: Plasma Lorlatinib Metabolite AUC24 at Steady State
Description: AUC24 was defined as area under the plasma concentration time profile during one dosing interval (24 hours).
Time Frame: Cycle 2 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
ng*hr/mL | NA (NA) — No PK parameter estimation was performed for the 1 treated participant

14. Secondary Outcome: Plasma Lorlatinib Metabolite AUClast After Single Dose
Description: AUClast was defined as area under the plasma concentration time profile from time 0 to the time of Clast.
Time Frame: Cycle 1 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
ng*hr/mL | NA (NA) — No PK parameter estimation was performed for the 1 treated participant

15. Secondary Outcome: Plasma Lorlatinib Metabolite AUClast at Steady State
Description: AUClast was defined as area under the plasma concentration time profile from time 0 to the time of Clast.
Time Frame: Cycle 2 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
ng*hr/mL | NA (NA) — No PK parameter estimation was performed for the 1 treated participant

16. Secondary Outcome: Plasma Lorlatinib Metabolite Cmax After Single Dose
Description: Cmax was defined as maximum plasma concentration and was observed directly from data.
Time Frame: Cycle 2 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
ng/mL | NA (NA) — No PK parameter estimation was performed for the 1 treated participant.

17. Secondary Outcome: Plasma Lorlatinib Metabolite Cmax at Steady State
Description: Cmax was defined as maximum plasma concentration and was observed directly from data.
Time Frame: Cycle 2 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
ng/mL | NA (NA) — No PK parameter estimation was performed for the 1 treated participant.

18. Secondary Outcome: Plasma Lorlatinib Metabolite Tlast After Single Dose
Description: Tlast was defined as the time of the last quantifiable concentration.
Time Frame: Cycle 1 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
hour | NA [NA to NA] — No PK parameter estimation was performed for the 1 treated participant.

19. Secondary Outcome: Plasma Lorlatinib Metabolite Tlast at Steady State
Description: Tlast was defined as the time of the last quantifiable concentration.
Time Frame: Cycle 2 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
hour | NA [NA to NA] — No PK parameter estimation was performed for the 1 treated participant

20. Secondary Outcome: Metabolite Ratio of Lorlatinib Metabolite for AUC24 (MRAUC24) at Steady State on Cycle 2 Day 1
Description: MRAUC24 was defined as metabolite ratio of lorlatinib metabolite for AUC24.
Time Frame: Cycle 2 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
Ratio | NA (NA) — No PK parameter estimation was performed for the 1 treated participant.

21. Secondary Outcome: Metabolite Ratio of Lorlatinib Metabolite for AUClast (MRAUClast) at Steady State on Cycle 2 Day 1
Description: MRAUClast was defined as metabolite ratio of lorlatinib metabolite for AUClast.
Time Frame: Cycle 2 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
Ratio | NA (NA) — No PK parameter estimation was performed for the 1 treated participant.

22. Secondary Outcome: Metabolite Ratio of Lorlatinib Metabolite for Cmax (MRCmax) at Steady State on Cycle 2 Day 1
Description: MRCmax was defined as metabolite ratio of lorlatinib metabolite for AUClast.
Time Frame: Cycle 2 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
Ratio | NA (NA) — No PK parameter estimation was performed for the 1 treated participant.

23. Secondary Outcome: Metabolite Ratio of Lorlatinib Metabolite for AUClast (MRAUClast) at Steady State on Cycle 1 Day 1
Description: MRAUClast was defined as metabolite ratio of lorlatinib metabolite for AUClast.
Time Frame: Cycle 1 day 1 at times 0 (predose), 0.5, 1, 2, 4, 6, 10, and 24 hours post lorlatinib dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Group B Mild Hepatic Impairment
Number analyzed (Participants) | 1
Ratio | NA (NA) — No PK parameter estimation was performed for the 1 treated participant.

ADVERSE EVENTS:
Time Frame: From Screening (within 28 days prior to Cycle 1 Day 1) through and including at least 28 days after after the last lorlatinib dose. The duration is approximately 42 days.
Description: AE information were reported by using the System Organ Class instead of preferred term to avoid the risk of re-identification of the participant.
Arm/Group | Group B Mild Hepatic Impairment
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group B Mild Hepatic Impairment (N=1)
Nervous system disorders (Nervous system disorders) | 1
Psychiatric disorders (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group B Mild Hepatic Impairment (N=1)
General disorders (General disorders) | 1
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1
Nervous system disorders (Nervous system disorders) | 1
Psychiatric disorders (Psychiatric disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to difficulties with enrolling eligible patients. Only 1 participant was enrolled in this study. Outcome measures and AE data were not reported as planned in the protocol because doing so would risk re-dentification of the individual participant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT03726333/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT03726333/SAP_001.pdf